CLINICAL TRIAL: NCT01591200
Title: A Parallel Group Randomized Open Blinded End Point Evaluation, Multicentric, Dose Escalation, Phase -II Study Assessing the Safety and Efficacy of Intraarterial (Hepatic) Ex-vivo Cultured Adult Allogenic Mesenchymal Stem Cells in Patients With Alcoholic Liver Cirrhosis
Brief Title: Dose Finding Study to Assess Safety and Efficacy of Stem Cells in Liver Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stempeutics Research Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRPL/LC/09-10/001
Record Dates: First submitted 2012-04-15; First posted 2012-05-03 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Alcoholic Liver Cirrhosis
Keywords: Alcoholic; Liver; Cirrhosis; Stem; Cells
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (No Intervention): This arm will receive standard protocol of care alone
- Stem cells high dose (Experimental): This arm will receive high dose of Allogeneic Mesenchymal Stem Cells
  Interventions: Biological: Allogeneic Mesenchymal Stem Cells
- Stem cells intermediate dose (Experimental): This arm will receive intermediate dose of Allogeneic Mesenchymal Stem Cells
  Interventions: Biological: Allogeneic Mesenchymal Stem Cells
- Stem cells low dose (Experimental): This arm will receive low dose of Allogeneic Mesenchymal Stem Cells
  Interventions: Biological: Allogeneic Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Stem Cells — High dose of Bone Marrow Derived Allogeneic Mesenchymal Stem Cells will be administered through the hepatic artery
  Arms: Stem cells high dose
Biological: Allogeneic Mesenchymal Stem Cells — Intermediate dose of Bone Marrow Derived Allogeneic Mesenchymal Stem Cells will be administered through the hepatic artery
  Arms: Stem cells intermediate dose
Biological: Allogeneic Mesenchymal Stem Cells — Low dose of Bone Marrow Derived Allogeneic Mesenchymal Stem Cells will be administered through the hepatic artery
  Arms: Stem cells low dose

SUMMARY:
This study will evaluate the safety and efficacy of mesenchymal stem cells in patients with cirrhosis of liver. Stem cells will be injected into the hepatic artery. Improvement in various parameters will be observed over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic cirrhotics between 18-65 years of age (diagnosed by clinical, biochemical, sonographic, radiological [CT scan] or histological evidence of cirrhosis and portal hypertension).
* Evidence of decompensated liver disease at screening (e.g. Child class B or C, Child-Pugh scores of ≥7 and <14).
* MELD scores of at least 10 (UNOS Meld calculator).
* Normal AFP Level
* Hb>10gm/dl.
* Female patients of childbearing age must be willing to use accepted methods of contraception during the course of the study
* Signed informed consent.

Exclusion Criteria:

* Patients likely to undergo liver transplantation during the duration of the study.
* Presence of advanced hepatic encephalopathy Grades 3 & 4 (West Haven criteria for grading of hepatic encephalopathy) at the time of screening
* Active variceal bleed.
* Refractory ascites.
* Evidences of autoimmune liver disease- ANA or Anti-LKM positivity.
* Platelet count < 30,000/mm3.
* Serum Sodium <129mEq/L.
* Serum Creatinine > 2 mg/dl.
* Hepatocellular carcinoma or other malignancies
* Active infectious disease.
* Presence of severe underlying cardiac, pulmonary or renal disease.
* Excessive alcohol (>30 gm of alcohol/day) use in the last 3 months before screening.
* Positive HbSAg or antibodies to HIV or HCV.
* Pregnancy or lactation.
* Participation in other clinical trials.
* Unwilling/unable to sign the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety | 2 years
  The type of adverse events, number of adverse events and proportion of patients with adverse events

SECONDARY OUTCOMES:
Liver function tests. | 2 years
  To assess the improvement in liver function
CT scan of abdomen. | 2 years
  To assess the improvement in liver structure
Change in MELD score | 2 years
  To assess the clinical improvement
Improvement in quality of life as assessed by SF 36 questionnaire | 2 years
  To assess the improvement in quality of life
Histological evaluation of liver biopsy by immunohistochemical staining for AFP, PCNA, SMA | 6 Months
  To assess the improvement in histopathology
Change in Child-Pugh score | 2 years
  To assess clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Dr. BV Tantry, MD., DM, Principal Investigator — KMC, Mangalore; Dr. Samir Shah, MD., DM, Principal Investigator — Breach Candy Hospital, Mumbai; Dr. Dinesh Kini, MD., DM, Principal Investigator — Manipal Hospital, India; Dr.Deepak N Amarapuraka, MD., DM, Principal Investigator — Bombay Hospital & Medical Research Center, Mumbai; Dr. VA Saraswat, MD., DM, Principal Investigator — SGPGI, Kucknow; Dr. Aejaz Habeeb, MD., DM, Principal Investigator — Centre for Liver Research & Diagnostics, Hyderabad; Dr Uma Devi, MD, Principal Investigator — Mediciti Hospital; Dr Sanjay Kolte Kolte, DNB., FCPS, Principal Investigator — Sahyadri Speciality Hospital; Dr Sandeep Nijhwan Nijhwan, MD., DM, Principal Investigator — SMS Medical College and Hospital; Dr. Nitin Pai, MD., DM, Principal Investigator — Ruby Hall clinic
Locations (10):
- India (10):
  - Centre for Liver Research & Diagnostics, Hyderabad, Andhra Pradesh
  - Mediciti Hospital, Hyderabad, Andhra Pradesh
  - Manipal Hospital, Bangalore, Karnataka
  - KMC Hospital, Mangalore, Karnataka
  - Institute of liver disease, HPB surgery and transplant Global Hospitals, Mumbai, Maharashtra
  - Bombay Hospital & Medical Research Center, Mumbai, Maharashtra
  - Ruby Hall clinic, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - SMS Medical college and Hospital, Jaipur, Rajasthan
  - SGPGI Lucknow, Lucknow, Uttar Pradesh